CLINICAL TRIAL: NCT00360126
Title: An Open-Label Extension Study to Assess the Safety of Lamotrigine in Subjects With Bipolar Disorder, Who Are in Remission Following a Manic/Hypomanic Index Episode or a Depressive Index Episode.
Brief Title: An Open-Label Extension Study Of Lamotrigine In Subjects With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA104753
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Bipolar Disorder
Keywords: Lamictal; lamotrigine; Open-Label Extension Study; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
The precursor study (SCA101469) was an open-label, prospective multicentre study in adult subjects diagnosed with bipolar disorder consisting of 36 weeks treatment with lamotrigine. The current study is to provide 12 months post study access to open-label lamotrigine for participants of the SCA101469 study.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* completed 32 weeks of open label treatment in study SCA101469 and, in the investigators opinion, has responded to lamotrigine therapy
* male or female subject

A female is eligible to enter and participate in this study if she is of:

1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or sterilised) or,
2. child-bearing potential, has a negative urine pregnancy test at screening, and agrees to one of the following contraceptive methods:

   * Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for a time interval after completion of premature discontinuation from the study to account for elimination of the investigational drug (a minimum of 5 half-lives or longer if the pharmacodynamic profile of the investigational drug warrants a longer time period); or,
   * Sterilisation of male partner; or,
   * Implants of levonorgestrel; or,
   * Injectable progestogen; or,
   * Oral contraceptive (combined or progestogen only); or,
   * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or,
   * Any other methods with published data showing that the lowest expected failure rate for that method is less than 1% per year; or,
   * Barrier method only if used in combination with any of the above acceptable methods.

     * willing and able to give written informed consent to participate in the study.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* subject experienced a 'mood episode' during participation in study SCA101469, or since completing participation in study SCA101469.
* participation in a clinical drug trial other than SCA101469 within the past 30 days or previous participation in this clinical study
* known hypersensitivity to lamotrigine
* in the investigator's judgement, the subject poses a current serious suicidal or homicidal risk, or has made a suicide attempt within the past 6 months.
* combination of carbamazepine and valproate
* concurrent lamotrigine therapy, other than that commenced in study SCA101469
* current or history of substance abuse
* diagnosis of epilepsy
* diagnosis or history of an obsessive-compulsive disorder, social phobia, or eating disorder
* significant cardiac, renal, cerebrovascular, or hepatic condition; no significant abnormalities in the laboratory tests or ECG recording performed during study SCA101469.
* unable to understand or implement instructions
* unresolved drug related adverse event or serious adverse event occurring in study SCA101469

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Australia (3):
  - GSK Investigational Site, Greenwich, New South Wales
  - GSK Investigational Site, Everton Park, Queensland
  - GSK Investigational Site, New Farm, Queensland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 participants were enrolled and randomized from 13 October 2005 to 12 February 2007.
Pre-assignment Details: Participants who had completed 32 weeks treatment period in study SCA101469 were enrolled in this extension study.
Groups:
- Lamotrigine: Participants received Lamotrigine tablets orally once daily up to 52 weeks in evenings or mornings (in case of non-tolerance) or the dose was administered twice daily if the morning dose was not tolerated.
Period: Overall Study
Arm/Group | Lamotrigine
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lamotrigine
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.64 (3.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: Participants]
  Australia | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event is therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Only SAEs were recorded and reported in this extension study.
Time Frame: Up to 54 weeks
Population: All subject population consisted of all participants enrolled into the study and received study drug.
Measure: Number; unit: Participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: SAEs were collected for 'All subject population'. Only SAEs were recorded and reported in this extension study. Other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.